CLINICAL TRIAL: NCT02032394
Title: Comparison of the Effect of Applying Povidone-iodine and Chlorhexidine Solutions for Perinea Washing on Bacteriuria Rate and Type in Patients With Urinary Catheter in Intensive Care Unit
Brief Title: Effect of Chlorhexidine on Bacteriuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Seyedreza Mazloum, Faculty member of Medical Surgical Nursing Department, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MUMS910212
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Urinary Tract Infection; Nosocomial Infection; Bacteriuria
Keywords: Chlorhexidine; Povidone-iodine; bacteriuria; Urinary Catheterization; Urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections; Cross Infection; Bacteriuria | interventions — Povidone-Iodine; Chlorhexidine; chlorhexidine gluconate; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine (Experimental): Washing of perineal area and proximal first 5 centimeters of catheter from mea, done by 15 ml of Chlorhexidine 0.2%, 3 times a day for 10 days.
  Interventions: Drug: Chlorhexidine
- Povidone-Iodine (Experimental): Washing of perineal area and proximal first 5 centimeters of catheter from mea, done by 15 ml of Povidone-iodine 10%, 3 times a day for 10 days.
  Interventions: Drug: Povidone-iodine
- Normal saline (Active Comparator): Washing of perineal area and proximal first 5 centimeters of catheter from mea, done by 15 ml of Normal saline 0.9%, 3 times a day for 10 days.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Povidone-iodine — 15 ml 10%, 3 imes a day for 10 days /external use for Washing perinea area and catheter first 5 centimeters
  Other Names: Betadine
  Arms: Povidone-Iodine
Drug: Chlorhexidine — 15 ml .2%, 3 imes a day for 10 days /external use for Washing perinea area and catheter first 5 centimeters
  Other Names: CHLORHEXIDINE GLUCONATE
  Arms: Chlorhexidine
Drug: Normal saline — 15 ml .9%, 3 imes a day for 10 days /external use for Washing perinea area and catheter first 5 centimeters
  Other Names: Chloride Sodium
  Arms: Normal saline

SUMMARY:
This study is conducted to determine and compare the effect of applying Povidone-iodine and Chlorhexidine solutions for perinea washing on bacteriuria rate and type in patients with urinary catheter in intensive care unit.

DETAILED DESCRIPTION:
This is a double blind randomized study with control group. The population is patients in intensive care unit of Shahid Beheshti hospital of Babol city. Main include criteria are 18-55 years old, need to having urine catheter for 10 days at least and no urinary infection in catheterization time. Main exclude criteria are appearing genital wound, allergic or dermatitis disorders. Sample size include 105 patients dividing in three equal groups of Povidone-iodine, Chlorhexidine and Normal saline randomly. Interventions are Washing perinea area and catheter first 5 centimeters by 15 ml of Povidone-iodine 10%, Chlorhexidine .2% or Normal saline .9%, 3 times a day for 10 days. Urine analysis are performed in days 1,3,5,7 and 9 after catheterization and urine cultures are performed in days 5 and 10 after catheterization for detection of bacteriuria and microorganism type.

ELIGIBILITY:
Inclusion Criteria:

* Must need a urinary catheter for 10 days at least
* Must have 18-55 years old
* Men subjects must doing circumcision already
* Urinary catheter must be apply in a standard method by researcher or via her supervision

Exclusion Criteria:

* No more tendency of patient or his/her significant other for continuing study
* Malignant disease such as prostate or uterine cancer
* History of recurrent urinary infection
* Congenital urinary system disorders
* history of allergy
* Immunodeficiency disorders
* Urinary system intervention in past sixth months
* Urinary infection at study start
* Positive urine analysis or urine culture results in first 3 days of study
* Abdominal or pelvic surgery
* Women having period during study
* Any allergic reaction or dermatitis resulted from applying study solutions
* Appearing genital wounds
* Diabetes mellitus
* Wound in genital area
* Discharging, transferring or dying in first week of study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Bacteriuria day 1 | day 1 after urinary catheterizatiion
  Bacteriuria is assessed according to result of urine analysis and is presented as positive or negative.
Bacteriuria day 3 | Day 3 after catheterization
  Bacteriuria is assessed according to result of urine analysis and is presented as positive or negative.
Bacteriuria day 5 | day 5 after catheterization
  Bacteriuria is assessed according to result of urine analysis and is presented as positive or negative.
Bacteriuria day 7 | Day 7 after catheterization
  Bacteriuria is assessed according to result of urine analysis and is presented as positive or negative.
Bacteriuria day 9 | Day 9 after cathetrization
  Bacteriuria is assessed according to result of urine analysis and is presented as positive or negative.

SECONDARY OUTCOMES:
Microorganism Type day 5 | Days 5 after catheterization
  Microorganism type is assessed according to result of Urine culture and is presented as the name of microorganism causing urinary infection.
Microorganism type day 10 | Day 10 after catheterization
  Microorganism type is assessed according to result of Urine culture and is presented as the name of microorganism causing urinary infection.

CONTACTS AND LOCATIONS:
Overall Officials: Seyedreza Mazloum, Ph.D., Study Chair — Medical Surgical Nursing Department, Mashhad University of Medical Sciences; Kamran Mohammadnia, Ms., Study Director — Postgraduate Department, Mashhad University of Medical Sciences; Tayyebe Pourghaznein, Ms., Study Director — Medical Surgical Nursing Department, Mashhad University of Medical Sciences; Ebrahim Alijanpoor, Specialist, Study Director — Anesthesia Department, Babol University of medical scienses
Locations (1):
- Shahid Beheshti Hospital, Babol, Mazandaran, Iran